CLINICAL TRIAL: NCT04121312
Title: Engaging Primary Care Patients in Online Weight Management Tools: A Pilot Study
Brief Title: Engaging Patients in Weight Loss Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201902013; OCR26064 (Other: UF OnCore)
Record Dates: First submitted 2019-10-03; First posted 2019-10-09 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facilitation Intervention (Experimental): A brief, web-based facilitation guide (called "Weight Loss Your Way Kickoff Materials") that encourages initial and sustained engagement in online tracking and social network tools for weight loss.The intervention also includes 8 emails sent over 12 weeks to further motivate use of the online tools and weight loss.
  Interventions: Behavioral: Facilitation Intervention

INTERVENTIONS:
Behavioral: Facilitation Intervention — See "arm" description

SUMMARY:
The overall aim of this study is to evaluate the acceptability and feasibility of a primary-care based approach to facilitating engagement in online behavior tracking and community support networks for weight loss ("facilitation condition") over 12 weeks among adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* PCPs:

  1. Employed as a PCP at a clinics in the UF health care system.
  2. Has practiced at current clinic for ≥1 year (self-report)
  3. Is employed ≥ 0.5 FTE (self-report)
  4. Has a patient panel that is majority adult (self-report)
* Patients: EHR-based criteria:

  1. Age 18-75
  2. Last BMI in EHR ≥30 kg/m2
  3. Has an appointment scheduled ("index appointment") with an enrolled primary care PCP 7-30 days after electronic data pull.
  4. Is enrolled in MyChart or has an email address in the IDR system.

     Self-report criteria:
  5. Self-reported BMI > 29 kg/m2 (to account for under-reporting)
  6. Response yes to question: "Would you be interested in learning strategies to help you lose weight?"
  7. Ability to read and understand English without assistance.
  8. Has either (a) a phone or tablet with a data plan OR (b) reliable access to Wi-Fi (via computer, phone or tablet) in their home.

Exclusion Criteria:

* PCPs:

  1. Planning to move out of the Gainesville or Jacksonville area in the next 12 months.
* Patients:

  1. Currently enrolled in formal weight loss program or a research study focused on changing diet, physical activity, or weight.
  2. In past month, has tracked the majority of their food intake on an app, website, or paper log an average of 3 or more days per week.
  3. Self-reported to be pregnant, breastfeeding, or planning to become pregnant in next 6 months.
  4. Currently undergoing radiation or chemotherapy for cancer.
  5. Self-reported cardiac event in past 6 months.
  6. Self-reported Heart Failure (also known as chronic heart failure or CHF).
  7. Planning to move out of the Gainesville or Jacksonville area (depending on which clinic they are recruited from) in the next 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Patient retention | 12 weeks
  Percent of enrolled patients completing the 12-week follow-up assessment. (NOTE: this is a feasibility pilot and is not conceptualized as having a single primary outcome)

SECONDARY OUTCOMES:
Provider retention | 4-6 months (depends on patient recruitment rate)
  Percent of enrolled providers who complete telephone interview at end of study
Percent of contacted providers who enroll | NA (depends on period of recruitment, approx 1 month)
  Percent of PCPs offered the study who consent
Percent of patients who enroll | NA (depends on period of recruitment, approx 2-4 months)
  Percent of patients contacted who are eligible and agree to participate.
Rate of patient recruitment | up to 16 weeks
  Patients recruited per month during active recruitment periods
Acceptability of intervention- provider | At end of intervention (about 4-6 months after start, depending on recruitment rate)
  Response to 5 study specific questions asking about alignment with priorities, fit in workflow, feasibility, perception of patient benefit, and time. Also, response to open ended question about acceptability.
Acceptability of intervention- patient: 12 study specific questions | 12 weeks
  Response to 12 study specific questions asking about experience with "Weight Loss Your Way" kickoff materials; open ended response to questions about acceptability of intervention during qualitative interviews (of portion of enrollees)
Initial engagement in Tracking tool and social network | 12 weeks
  Portion of patients who initially engage with tracking tool (i.e., log at least one food item or physical activity) and with social network (i.e., who report reading message board or posting at least once) (tracking and social network examined separately)
Sustained engagement in Tracking tool and social network | 12 week assessment (queried about prior week)
  Portion of patients who have used the tracking tool and social network at least once in past week at 12 week assessment (tracking and social network examined separately)
Weight change | baseline to 12 weeks
  Mean weight loss (kgs) and portion of participants achieving 3% body weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Megan McVay, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health at the University of Florida, Gainesville, Florida
  - UF Health - Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No